CLINICAL TRIAL: NCT06015724
Title: A Phase 2 Study Evaluating the Efficacy of Anti-CD38 Antibody in Combination With KRAS Vaccine and Anti-PD-1 Antibody in Subjects With Pancreatic Ductal Adenocarcinoma and Refractory Non-Small Cell Lung Cancer
Brief Title: Anti-CD38 Antibody With KRAS Vaccine and Anti-PD-1 Antibody in Subjects With Pancreatic Ductal Adenocarcinoma and Refractory Non-Small Cell Lung Cancer
Acronym: DARANIVOVAX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Bristol-Myers Squibb (Industry); Janssen, LP (Industry); Targovax ASA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005625
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Refractory Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — daratumumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pancreatic Ductal Adenocarcinoma (Experimental)
  Interventions: Drug: Daratumumab; Biological: KRAS vaccine; Drug: Nivolumab
- Refractory Non-Small Cell Lung Cancer (Experimental)
  Interventions: Drug: Daratumumab; Biological: KRAS vaccine; Drug: Nivolumab

INTERVENTIONS:
Drug: Daratumumab — anti-CD38 monoclonal antibody (mAb)
  Other Names: Darzalex Faspro
Biological: KRAS vaccine — Stimulon QS-21 and Targovax TG01
Drug: Nivolumab — anti-PD-1 (programmed cell death protein 1) monoclonal antibody (mAb)
  Other Names: BMS-936558

SUMMARY:
The goal of this clinical trial is to test the safety and tolerability of anti-CD38 monoclonal antibody (mAb), daratumumab, in combination with KRAS vaccine (Targovax TG-01/Stimulon QS-21) when given with anti-PD-1 (programmed cell death protein 1) mAb (nivolumab) in patients with advanced non-small cell lung cancer (NSCLC) or pancreatic ductal adenocarcinoma (PDAC). The main questions it aims to answer are:

* How well does daratumumab and nivolumab, when given with a vaccine, control or stop these types of cancer?
* How well does participants bodies handle these study drugs?
* Does this combination of study drugs help participants live longer? Participants will receive daratumumab, nivolumab with KRAS vaccine and have regular tests and procedures to follow how the participants are doing on these study drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Patients with advanced NSCLC, progressing on frontline anti-PD-1/PD-L1 containing therapy (patient with rapid tumor progression will be excluded) and PDAC patients who failed one prior treatment.
3. Measurable disease as defined by irRECIST criteria (See Section 7) NOTE: Tumor lesions in a previously irradiated area are not considered measurable disease; Disease that is measurable by physical examination only is not eligible.
4. All patients with mutant KRAS status in either codon 12 (12A, C, D, R, S, V) or 13 (13D) will be included. The status of KRAS and LKB1 will be determined. For patients with KRAS G12C-mutated NSCLC, prior treatment with G12C-targeted therapy will be allowed; a wash-out period of 1 week from the last administration of targeted therapy would be allowed.
5. Prior treatment:

   * For NSCLC: Anti-PD1/PD-L1 containing therapy; a wash-out period of 4 weeks from the last administration of therapy would be allowed.
   * For PDAC: Patients who failed one prior treatment.
6. Provide written informed consent.
7. Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study).
8. Willingness to provide mandatory blood specimens for correlative research.
9. Willingness to provide mandatory tissue specimens for correlative research.
10. ECOG Performance Status (PS) 0, 1 or 2.
11. The following laboratory values obtained ≤14 days prior to registration:

    * Hemoglobin ≥9.0 g/dL
    * Absolute neutrophil count (ANC) ≥1500/mm3
    * Platelet count ≥100,000/mm3
    * Total bilirubin ≤1.5 x ULN (upper limit of normal)
    * ALT and AST ≤3 x ULN (≤5 x ULN for patients with liver involvement)
    * PT (prothrombin time)/INR/aPTT (activated partial thromboplastin time) ≤1.5 x ULN OR if patient is receiving anticoagulant therapy and INR or aPTT is within target range of therapy
    * Calculated creatinine clearance (CrCl) ≥20 mL/min using the Cockcroft-Gault formula
12. Negative pregnancy test done ≤7 days prior to registration, for persons of childbearing potential only.

Exclusion Criteria:

1. Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

   * Pregnant persons
   * Nursing persons
   * Persons of childbearing potential who are unwilling to employ adequate contraception
2. Any of the following prior therapies:

   * Daratumumab or other anti-CD38 therapies
   * Surgery ≤3 weeks prior to registration
   * Chemotherapy ≤4 weeks prior to registration
   * For NSCLC: anti-PD-1/PD-L1 therapy or second line therapy ≤4 weeks prior to registration; for PDAC: Prior treatment with an anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T cell co-stimulation or checkpoint pathways.
   * Focal radiation therapy within 14 days prior to first study treatment with the exception of palliative radiotherapy for symptomatic management but not on measurable extramedullary plasmacytoma. Participants must have recovered (ie, Grade ≤1 or at baseline) from radiation-related toxicities prior to first study treatment.
   * Treatment with complementary medications (e.g., herbal supplements or traditional Chinese medicines) to treat the disease under study within <2 weeks prior to first study treatment. Such medications are permitted if they are used as supportive care.
   * Treatment with any live / attenuated vaccine within 30 days of first study treatment.
3. Co-morbid systemic illnesses or other severe concurrent disease, which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
4. Uncontrolled intercurrent illness including, but not limited to:

   • Ongoing or active infection

   • Symptomatic CHF (class II and above that are not properly controlled on maintenance therapy or that have been hospitalized in the last 4 weeks for heart failure)
   * Unstable angina pectoris
   * Cardiac arrhythmia
   * Or psychiatric illness/social situations that would limit compliance with study requirements.
5. Receiving any other investigational agent, which would be considered as a treatment for the primary neoplasm.
6. Other active malignancy ≤5 years prior to registration. EXCEPTIONS: Squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix or breast, or other non-invasive lesions that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 3 years.
7. History of myocardial infarction ≤6 months, or CHF (class II and above that are not properly controlled on maintenance therapy or that have been hospitalized in the last 4 weeks for heart failure) requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias.
8. Patients with known primary CNS malignancy or symptomatic CNS metastases are excluded, with the following exceptions:

   * Patients with asymptomatic untreated CNS disease may be enrolled, provided all of the following criteria are met:

     o Evaluable or measurable disease outside the CNS

     o No metastases to brain stem, midbrain, pons, medulla, cerebellum, or within 10 mm of the optic apparatus (optic nerves and chiasm)

     o No history of intracranial hemorrhage or spinal cord hemorrhage

     o No ongoing requirement for dexamethasone for CNS disease; patients on a stable dose of anticonvulsants are permitted.

     o No neurosurgical resection or brain biopsy ≤28 days prior to registration
   * Patients with asymptomatic treated CNS metastases may be enrolled, provided all the criteria listed above are met as well as the following:

     * Radiographic demonstration of improvement upon the completion of CNS-directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study
     * No stereotactic radiation or whole-brain radiation ≤28 days prior to registration
     * Screening CNS radiographic study ≥4 weeks from completion of radiotherapy and ≥ 2 weeks from discontinuation of corticosteroids
9. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins or vaccines.
10. Patients with a plan to receive yellow fever or other live (attenuated) vaccines during the course of study.
11. Patients who have a history or current evidence of bleeding disorder, i.e., any hemorrhage/bleeding event of CTCAE Grade ≥2, ≤28 days prior to registration.
12. Patients on supraphysiologic doses of steroids taken within 6 weeks of study drug initiation. Exceptions:

    a) Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after PI confirmation has been obtained.

    b) Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.

    c) Patients who received a brief taper of corticosteroids (< 4 weeks duration) (exceeding 10mg daily prednisone or equivalent) are eligible upon PI confirmation.

    d) Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
13. Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease.
14. History or risk of autoimmune disease, including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis. Note: Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone are eligible. Patients with controlled Type 1 diabetes mellitus (T1DM) on a stable insulin regimen are eligible. Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

    o Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations

    o Rash must cover less than 10% of body surface area (BSA)

    o Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, flucinolone 0.01%, desonide 0.05%, aclometasone dipropionate 0.05%)

    o No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids).
15. History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest CT scan. Note: History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
16. Any infection > Grade 2 ≤4 weeks prior to registration, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
17. Subject is

    * Seropositive for HIV.
    * Seropositive for hepatitis B (defined by a positive test for HBsAg). Subjects with resolved infection (i.e., subjects who are HBsAg negative but positive for anti-HBc and/or anti-HBs) must be screened using RT-PCR measurement of HBV DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
    * Seropositive for hepatitis C (except in the setting of a SVR, defined as aviremia at least 12 weeks after completion of antiviral therapy).
    * Note: HIV and HCV testing at screening is at the investigator's discretion. Serological testing if already performed within 3 months of starting the study drugs may be used. All subjects will be tested locally for HBsAg, Anti-HBs, and Anti-HBc at Screening.

19. COPD with a FEV1 < 50% of predicted normal. Note that FEV1 testing is required for participants suspected of having COPD and participants must be excluded if FEV1 is < 50% of predicted normal.

20. Moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification. Note that participants who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate.

21. Prisoners or subjects who are compulsory detained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) (Efficacy) | every 8 weeks, approximately 2 years
  Evaluation of response by ORR by irRECIST criteria. Response classification will follow the irRECIST criteria and will be defined as PR or CR. Patients who are lost to follow-up without a valid response assessment will be classified as NR (non-responder, progression). The ORR will be computed for all patients with at least one cycle of the study drug.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From start of intervention until 30 days following discontinuation of intervention, approximately 2 years
  Incidence rate of Adverse Events
Progression Free Survival (PFS) | at 6 months and 9 months
  PFS will be defined as the time in days from study entry until progression or death.
Duration of Response (DOR) | approximately 3 years
  DoR is defined as the length of time tumor continues to respond to the treatment.
Clinical Benefit Rate (CBR) | approximately 2 years
  CBR classification will follow the irRECIST criteria and will be defined as the percentage of patients who achieved stable disease (SD) or better response.
Overall Survival | approximately 3 years
  OS will be defined as the time in days from study entry until death. All events of death will be included, regardless of whether the event occurred while the subject was still taking study drug, or after the subject discontinued study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Samir Khleif, MD, Principal Investigator — Georgetown University
Locations (2):
- United States (2):
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No